CLINICAL TRIAL: NCT06363578
Title: Comparing the Analgesic Effects of Different Doses of Dexmedetomidine as an Adjuvant in External Oblique Intercostal Plane Block in Splenectomy: A Randomized Trial
Brief Title: Different Doses of Dexmedetomidine in External Oblique Intercostal Plane Block in Splenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR604/3/24
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Dexmedetomidine; External Oblique Intercostal Plane Block; Splenectomy
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group dexmedetomidine 0.5 (Experimental): Patients will receive 29 ml bupivacaine 0.25% + 1 ml dexmedetomidine 0.5 μg/kg diluted in saline.
  Interventions: Drug: Dexmedetomidine 0.5 μg/kg
- Group dexmedetomidine1 (Experimental): Patients will receive 29 ml bupivacaine 0.25% + 1 ml dexmedetomidine 1 μg/kg diluted in saline.
  Interventions: Drug: Dexmedetomidine 1 μg/kg

INTERVENTIONS:
Drug: Dexmedetomidine 0.5 μg/kg — Patients will receive 29 ml bupivacaine 0.25% + 1 ml dexmedetomidine 0.5 μg/kg diluted in saline.
  Arms: Group dexmedetomidine 0.5
Drug: Dexmedetomidine 1 μg/kg — Patients will receive 29 ml bupivacaine 0.25% + 1 ml dexmedetomidine 1 μg/kg diluted in saline.
  Arms: Group dexmedetomidine1

SUMMARY:
The aim of this study is to compare the analgesic effects of different doses of dexmedetomidine as an adjuvant in external oblique intercostal plane block (EOIPB) in splenectomy.

DETAILED DESCRIPTION:
External oblique intercostal plane block (EOIPB) was reported by Elsharkawy et al . It is a novel block, which has been described as an important modification of the fascial plane blocks that can consistently involve the upper lateral abdominal walls. In comparison to quadratus lumborum block (QLB) and erector spinae plane block (ESPB) , EOIPB has the benefit of being performed when the patient is supine. It also has an advantage over serratus intercostal plane block (SIPB) in that it produces greater analgesia throughout the midline of the abdomen.

Dexmedetomidine is used for sedation in patients admitted to the intensive care unit (ICU). Dexmedetomidine is a selective alpha 2- adrenoceptor agonist possessing sedative, anxiolytic, and analgesic properties without the development of respiratory depression . Several studies have shown that dexmedetomidine has an anesthetic sparing effect, which has led to its use as a general adjuvant for prolonging peripheral nerve block duration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status II-III.
* Scheduled for splenectomy.

Exclusion Criteria:

* Body mass index (BMI) ≥35 kg/m2
* History of abdominal surgery.
* Infection at the injection site.
* Drug abuse.
* Allergic reaction to local anesthetics.
* Coagulation abnormalities.
* Pregnancy.
* Severe cardiovascular problems.
* Diabetic neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 48 hour Postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4. NRS will be assessed at 0, 4, 8, 12, 18, 24, 36 and 48 h postoperatively.
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable").

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Total morphine consumption | 48 hour postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4. NRS will be assessed at 0, 4, 8, 12, 18, 24, 36 and 48 h postoperatively.
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable").
Degree of pain | 48 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable").
  Numerical rating Scale (NRS) will be assessed at 0, 4, 8, 12, 18, 24, 36 and 48 h postoperatively.
Heart rate | Till the end of surgery
  Heart rate will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Mean arterial pressure | Till the end of surgery
  Mean arterial pressure will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
The incidence of adverse events | 48 hour postoperatively
  Adverse events such as local anesthetic systemic toxicity (LAST), bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author